Official Title:

A Single Arm, Open Label Multicentre Extension Study of Bevacizumab in Patients With Solid Tumours on Study Treatment With Bevacizumab, at the End of A F. Hoffmann-La Roche and/or

Genentech Sponsored Study

NCT Number: NCT01588184

**Document Date:** SAP Version 3: 18-February-2019



Final version 3.0 / 18-FEB-2019

| | SPONSOR: ROCHE |
|------------------|------------------------|
| | PROTOCOL NUMBER: |
| | MO25757 |
| | TISTICAL ANALYSIS PLAN |
| Author: Version: | Final 3.0 |
| Date: | 18-FEB-2019 |



Final version 3.0 / 18-FEB-2019

# 1 Cover and signature pages

| Sponsor: | F.Hoffmann-La Roche Ltd |
|---|---|
| Protocol Number: | MO25757 |
| A Single Arm, Open Label Multicentre Extension St Bevacizumab in Patients with Solid Tumours on Study Tru with Bevacizumab, at the End of a F. Hoffmann-la Roche Genentech Sponsored Study | |
| Document Version No | Final v3.0 |

We, the undersigned, confirm that we have read, understood and agree to the content of this document and hereby authorise its approval.

| Name Title, Organisation | Signature | Date |
|--------------------------|-----------|------|



Final version 3.0 / 18-FEB-2019

| Sponsor: | F.Hoffmann-La Roche Ltd |
|---|---|
| Protocol Number: | MO25757 |
| Study Title: | A Single Arm, Open Label Multicentre Extension Study of Bevacizumab in Patients with Solid Tumours on Study Treatment with Bevacizumab, at the End of a F. Hoffmann-la Roche and/or Genentech Sponsored Study |
| Document Version No | Final v3.0 |

We, the undersigned, confirm that we have read, understood and agree to the content of this document and hereby authorise its approval.

| Name Title, Organisation | Signature | Date |
|--------------------------------|-----------|------|
| F.Hoffmann-La Roche Ltd | | |
| , MD. F.Hoffmann-La Roche Ltd | | |



Final version 3.0 / 18-FEB-2019

## **Table of Contents**

| 1 | Cover | Cover and signature pages | |
|---|---|---|---|
| 2 | List of | st of abbreviations 6 | |
| 3 | Introd | Introduction6 | |
| 4 | Study Objectives | | |
| 5 | Study | Design | 7 |
| | 5.1 | STUDY DESIGN AND POPULATION | 7 |
| | 5.2 | STUDY TREATMENTS AND ASSESSMENTS | 7 |
| | 5.3 | RANDOMIZATION AND BLINDING | 9 |
| | 5.4 | SAMPLE SIZE JUSTIFICATION | 9 |
| 6 | Statist | tical Considerations | 10 |
| 7 | Analys | sis Sets | 12 |
| 8 | Metho | ods of Analyses and Presentations | 13 |
| | 8.1 | SUBJECT DISPOSITION | 13 |
| | 8.2 | PROTOCOL DEVIATIONS AND/OR VIOLATIONS | 13 |
| | 8.3 | DEMOGRAPHIC AND BASELINE CHARACTERISTICS | 14 |
| | 8.4 | MEDICAL HISTORY | 14 |
| | 8.5 | PRIOR AND CONCOMITANT MEDICATION | 14 |
| | 8.6 | STUDY DRUG EXPOSURE AND/OR COMPLIANCE | 15 |
| | | 8.6.1 Bevacizumab Exposure | |
| | | 8.6.2 Non-IMP Exposure | |
| | 8.7 | EFFICACY DATA ENDPOINTS AND ANALYSES | |
| | | 8.7.2 Secondary Efficacy Endpoints and Analysis | |
| | 8.8 | PHARMACOKINETIC/ PHARMACODYNAMIC ENDPOINTS AND ANALYSES | |
| | 8.9 | QUALITY OF LIFE OR PHARMACOECONOMIC ENDPOINTS AND ANALYSES | |
| | 8.10 | SAFETY DATA ENDPOINTS AND ANALYSES | 18 |
| | | 8.10.1 Adverse Events (AEs) | 18 |
| | | 8.10.2 Vital signs | |
| | | 8.10.3 Other safety data | |
| 9 | | m Analyses | |
| 10 | Document History | | |
| 11 | References | | |
| 12 | Apper | ndices | 22 |
| | | B 4 (74 | 444/50 |



Final version 3.0 / 18-FEB-2019

12.1Tables, Figures and Listing shells2212.1.1In-text Tables, Figures and Listing shells2712.1.2EudraCT Tables3512.1.3Post-text Tables, Figures and Listing shells3812.2Imputation of partial dates74



Final version 3.0 / 18-FEB-2019

## 2 List of abbreviations

BC Breast Cancer
OC Ovarian Cancer
PC Peritoneal Carcinoma
CRC Colorectal Cancer
RCC Renal Cell Carcinoma

NSCLC Non-Squamous non-Small Cell Lung Cancer

GBM Glioblastoma SFU Safety Follow-up

PFS Progression free survival

OS Overall survival KM Kaplan Meir

SOC System Organ Class
PT Preferred Term
Bev. Bevacizumab
Treat. Treatment
AE Adverse Event

SAE Serious Adverse Event

AESI Adverse Event of Special Interest

MedDRA Medical Dictionary for Regulatory Activities

NCI CTC-AE National Cancer Institute Common Toxicity Criteria for Adverse Events

P-trial Parent trial E-trial Extension trial

PTAP Post-Trial Access Program

PDMS Protocol Deviation Management System
RECIST Response Evaluation Criteria in Solid Tumours

SAP Statistical analysis plan

## 3 Introduction

The purpose of this document is to describe the statistical methods, data derivations and data summaries to be employed in this Single Arm, Open Label Multicentre Extension Study of Bevacizumab in Patients with Solid Tumours on Study Treatment with Bevacizumab, at the End of a F. Hoffmann-la Roche and/or Genentech Sponsored Study.

The preparation of this statistical analysis plan (SAP) has been based on International Conference on Harmonisation (ICH) E3 and E9 Guidelines and in reference to Protocol MO25757 (version 3.0, 08Nov2018).

Template Author: Version 3.0 16AUG2017




Final version 3.0 / 18-FEB-2019

## 4 Study Objectives

**Primary objectives** of this study are as follows:

- To provide continued Bevacizumab therapy as single agent or in combination with an anti-cancer drug to patients with cancer who were previously enrolled in a Roche/Genentech sponsored Bevacizumab study (i.e. the Parent, P-trial) and who derived benefit from the therapy administered in the P-trial.
- To collect safety data with regard to long-term administration of Bevacizumab.

## 5 Study Design

#### 5.1 STUDY DESIGN AND POPULATION

This study is a multicenter, open-label, single-arm phase IIIb/IV trial in patients with solid tumours. The primary aim is to provide continued Bevacizumab therapy to cancer patients who benefit from the therapy administered in the P-trial until progression of their disease, therefore this is an open labelled, single arm, non-comparative study. Patients on Bevacizumab at study end of the P-trial should be enrolled immediately thereafter into this E-trial. Patients will receive treatment with Bevacizumab as during their P-trial until progression of disease, unacceptable toxicity, withdrawal of consent, death or transition to another option for treatment with bevacizumab (e.g. licensed product or Post-Trial Access Program [PTAP]) (whichever occurs first).

This study is a multi-national trial and the number of countries and centers is open. The number of patients to be enrolled over the planned recruitment period of approximately 5 years is open. This E-trial will end after the last patient safety follow-up (SFU) visit (latest 30 days after last patient permanently discontinues bevacizumab treatment in this E-trial).

#### **5.2 STUDY TREATMENTS AND ASSESSMENTS**

All patients must provide written informed consent before any E-trial-specific assessments or procedures are performed. Patients must fulfil all of the inclusion and none of the exclusion criteria to be enrolled in the E-trial.

Patients in this study will receive Bevacizumab at doses of 2.5 or 5 mg/kg/week every 2 or 3 weeks in line with the treatment schedule and dose as mandated by the P-trial, i.e.:

- Bevacizumab 7.5 or 15 mg/kg IV on day 1 every 3 weeks or
- Bevacizumab 5 or 10 mg/kg IV on day 1 every 2 weeks

The dose and schedule of Bevacizumab will be the same as during treatment in the P-trial.



Final version 3.0 / 18-FEB-2019

Treatment with Bevacizumab will be continued during the E-trial and will not be reduced for reasons other than a >10% change (loss or gain) in weight from baseline (at rollover assessment). Missed doses will not be administered subsequently. Treatment should not be omitted for more than 42 days unless because of planned surgery requiring bevacizumab interruption during P-trial. Bevacizumab can be restarted only after Sponsor's medical monitor approval.

At each cycle, Bevacizumab must be administered before concurrent anti-cancer therapy treatment at the same clinic visit, for oral agents the patients are allowed to follow their normal schedule.

Patients will receive treatment with Bevacizumab as during their P-trial until one of the following occurs:

- progression of disease;
- unacceptable Bevacizumab toxicity;
- withdrawal of consent;
- death;
- transition to another option for treatment with bevacizumab (e.g. licensed product).

The schedule of assessments is given in Table 1 below:

**Table 1.** Schedule of mandatory\* assessments

| | Roll over from P-<br>trial into E-Trial<br>(Day -14 to Day 1) | Treatment period Per cycle | Safety FU <sup>§</sup> |
|---|---|---|---|
| Informed Consent | X | | |
| Confirmation of eligibility | X | | |
| Patient characteristics | X | | |
| (Gender, date of birth, | | | |
| tumour type) | | | |
| Pregnancy test for WOCP# | X | | |
| Weight | | X | |
| Bevacizumab | | X+ | |
| Other P- trial anti-cancer | | | |
| IMP(s) if applicable** | | | |
| Progression assessment | | Per local | |
| | | standard° | |



Final version 3.0 / 18-FEB-2019

| AE | Х | Х | Х |
|---------------|---|---|---|
| Survival info | | Х | Х |

 $<sup>^{\</sup>S}$  (1) for patients who withdraw from the trial for reasons other than transition to another option for treatment with bevacizumab, 30 ( $\pm$  3) days after the last dose of bevacizumab (or other P-trial IMP(s), if applicable) and (2) for patients who withdraw from the trial to transition to another option for treatment with bevacizumab, before administration of non-trial bevacizumab outside of the study.

#### 5.3 RANDOMIZATION AND BLINDING

There will be no randomization or blinding to treatment as the study is a multicenter open label study. All patients in this study will receive Bevacizumab.

### **5.4 SAMPLE SIZE JUSTIFICATION**

This is an E-trial. Patients will be enrolled from qualifying P-trials. The formal estimation of sample size is not possible.

<u>Table 2</u> below presents a few possible scenarios for percentage of AEs grade  $\geq$  3 related to Bevacizumab with corresponding 95% Clopper-Pearson exact confidence intervals.

**Table 2.** Scenarios for Percentage and Number of Patients with AEs grade ≥ 3 related to Bevacizumab and corresponding Confidence Intervals

| Sample Size | Percentage and Number of<br>Patients with AEs grade ≥3<br>related to bevacizumab | 95% Clopper Pearson exact confidence interval |
|---|---|---|
| 50 | 10% (5 patients) | 3% - 22% |
| 50 | 20% (10 patients) | 10% - 34% |
| 100 | 10% (10 patients) | 5% - 18% |
| 100 | 20% (20 patients) | 13% - 29% |

It is difficult to estimate at this stage how many patients will be enrolled in this study. Assuming

<sup>#</sup> Pregnancy test: WOCP will have a serum pregnancy test no more than 7 days prior to the first trial treatment or no more than 14 days (with a confirmatory urine pregnancy test within 7 days prior to the first trial treatment).

<sup>\*</sup>Additional assessments (as per local standard and clinical judgement of the investigator) will only be documented in the patients' source documents

<sup>°</sup> The same method(s) as per P-trial are recommended

<sup>+ 1</sup>st Bevacizumab dose in MO25757 E-trial to be within 42 days of last dose in P-trial

<sup>\*\*</sup> classified as non-IMP in the E-trial



Final version 3.0 / 18-FEB-2019

a sample size of 100 patients then the percentage of patients with at least one AEs grade  $\geq$  3 related to Bevacizumab could be estimated to be within 5%-18% with a probability of 95% and assuming observed rate of patients with at least one AEs grade  $\geq$  3 of 10%.

The sample size was estimated using SAS Version 9.2 and nQuery Version 6.

## 6 Statistical Considerations

The following rules will be considered:

- Post-text Tables, Figures and Listings:
  - o Page Orientation: Landscape
  - o **Post-text outputs**, will be generated in .lst and converted to rtf.
  - o Font: Courier New font with minimum of 9 point font size
  - o Margins: top: 1", bottom: 0.8", left: 1.5" and right: 1.15" on A4 paper (i.e. line size of 120 and page size of 42)
- In-text Tables, Figures and Listings:
  - o Page Orientation: Portrait where possible
  - Post-text outputs, Report outputs (i.e. in-text outputs) will be generated using SAS ODS RTF with no borders or framing around table elements
  - o **Font**: Arial font with minimum of 9 point font size
- Columns header will be left aligned.
- Treatment labels: unless otherwise stated, all patients will be summarized under indication. Note a P-trial can be listed under more than one indication. The following labels will be used. Listing of P-trials with their indication can be found in section 12.2.
  - o BC
  - o OC or PC
  - o CRC
  - o RCC
  - o NSCLC
  - $\circ$  GBM
  - o Total
- Visit labels: the labels for the visits of the study are displayed in <u>Table 3</u>.
- Continuous variables (e.g., age) will be summarized using the number of observations (n), mean, standard deviation (SD), median, minimum, and maximum.



Final version 3.0 / 18-FEB-2019

- Categorical variables (e.g., sex, race) will be summarized using the number of observations (n) and percentage in each category.
  - The number of missing values will be presented as a separate category with no percentage, but only if 1 or more patients have missing data for the summary. Otherwise, all categories will be presented (even if no patients are counted in the category).
  - Counts of zero in any category will be presented without percentage.
     Precision for reporting derived endpoints will be determined by the statistician as appropriate for the study.
  - Except otherwise specified, percentages will be calculated based on the number of patients in the population

### • Precision of summary statistics:

- o Integer Sample size (n, N) and number of missing responses (if displayed)
- One additional decimal place than reported/collected mean, geometric mean, median, other percentile, confidence interval
- Two additional decimal places than reported/collected standard deviation
- o Same number of decimal places as reported/collected minimum, maximum
- Percentages –one decimal places
- All listings will be presented by Indication, P-trial, Non-IMP regimen, Country, Center/Patient and Age/Sex, and if applicable visit, assessment, assessment date/time and assessment (in order collected on CRF, unless specified otherwise).
- As Indication is not collected in the eCRF, for each P-trial the indication will be provided by Roche to be included in the analysis datasets.
- Summaries by P-trial should only be presented where there are at least 5 patients contributing from a P-trial.
- Study day calculations will be as follows. The calculation will result in dates prior to the date of first drug intake in the E-trial being presented as negative days, and those occurring on or after the date of first drug intake in the E-trial as Day 1 or later, i.e., there will be no Day 0.
  - o [date of interest date of first drug intake in the E-trial + 1] when the date of interest is on or after the date of first drug intake in the E-trial;
  - o [date of interest date of first drug intake in the E-trial] when the date of interest is prior to the date of first drug intake in the E-trial].
  - Missing if the patient was not treated in the E-trial.
- Days since last treatment (of Bevacizumab) in E-trial will be calculated to be presented in some TFLs, as mentioned in corresponding shells. The calculation is similar to the study day calculation:



Final version 3.0 / 18-FEB-2019

- o [date of interest date of last drug intake in the E-trial+1] when the date of interest is on or after the date of last drug intake in the E-trial;
- o [date of interest date of last drug intake in the E-trial] when the date of interest is prior to the date of last drug intake in the E-trial;
- Missing if the patient was not treated in the E-trial.
- Days since initial treatment (of Bevacizumab) in P-trial will be calculated to be presented in some TFLs, as mentioned in corresponding shells. The calculation is similar to the study day calculation and will result in positive days:
  - o [date of interest date of first drug intake in the P-trial+1]
- Dates will be presented in format DDMMMYYYY.
- Dictionary names and versions will be included in the footnotes of the adverse events tables and listings.
- The following partial dates will be imputed following the standard document, "Imputation Rules for Partial Dates" (see Section 12.3):
  - o Partial Adverse Event start and stop dates to determine the study days.

Table 3. Visit labels

| Visit Name | Visit Label for Tables | Visit Label for<br>Listings/Figures |
|---|---|---|
| Baseline (Day -14 to Day 1) | Baseline | BL |
| Treatment Period - Cycle x Day 1 to 14 | Cycle X | Cycle x |
| Treatment Period - Cycle x Day 1 to 21 | Cycle X | Cycle x |
| End of Treatment | End of Treatment | EoT |
| Safety Follow Up | Follow-Up | FU |
| End of Study | End of Study | EoS |

## 7 Analysis Sets

The following populations will be considered in the data analysis:

#### All patients population:

All patients population consists of all patients who are enrolled regardless of whether they received study drug only in the P-trial or not. This population will be used to summarize patient disposition, and major protocol deviations.



Final version 3.0 / 18-FEB-2019

## **Safety Population:**

The Safety population will include all enrolled patients in the E-trial who received at least one dose of Bevacizumab during this study. All drug exposure, compliance, efficacy and safety summaries and analyses will be presented for the safety population.

## **Methods of Analyses and Presentations**

#### 8.1 SUBJECT DISPOSITION

The number and percentage of patients enrolled, in the safety population and discontinued from Bevacizumab with corresponding reason for discontinuation will be summarized and listed by indication and overall. The frequency and percentages of reasons for patients who discontinued from the study will be tabulated by indication and overall. The number of patients in each analysis population will also be summarized similarly.

In addition, the median observation time, its 95% confidence interval and standard error as well as the 25% and 75% estimate of the observation time, the number of patients censored and with event will be summarized by indication and overall, using a reverse Kaplan-Meier. The observation time will be derived as follows:

If the patient completed the safety follow-up (i.e. safety follow-up visit performed), the observation time is calculated as follows:

Observation time (days) = (Date of safety follow-up visit - Date of first dose of Bevacizumab from E-trial) + 1.

If the patient has not completed the safety follow-up visit (for example the patient is lost-to follow-up, died or ongoing) then the patient will be censored at the last date of last known alive. Date of last known alive is the date of the last visit performed or if the patient died the day prior to the date of death.

Observation time (days) = (Date of last known alive - Date of first dose of Bevacizumab from E-trial) + 1.

The number of patients in each center, each P-trial and each indication, will be summarized overall to show the contribution of each P-trial and center to the E-trial. Supportive listing of Ptrial contribution and information will be provided.

### 8.2 PROTOCOL DEVIATIONS AND/OR VIOLATIONS

Non-compliance with the inclusion/exclusion criteria or major deviations from the protocol during the study conduct are considered protocol deviations. All protocol deviations will be recorded on the Roche Protocol Deviation Management System (PDMS) system and will be



Final version 3.0 / 18-FEB-2019

reviewed on an ongoing basis by a Medical Monitor and assigned a severity. Pre-defined rules and categories for protocol deviations have been defined at the beginning of the trial and are included in the PDMS. At the time of database lock all protocol deviations will be extracted from the PDMS system and reviewed for final approval. There will be one record per subject per protocol deviation. All protocol deviations will be listed by P-trial, country, center and patient.

The following major protocol deviations will be summarized:

- Inclusion criteria 2 (Patient is treated with bevacizumab at the end of the Roche/Genentech sponsored P-trial and continues to have benefit as judged by the investigator) and inclusion criteria 3 (Eligible for continuation of bevacizumab treatment at the end of the P-trial, according to P-trial protocol)
- Exclusion criteria 8 (Evidence of any AE potentially attributable to bevacizumab, for which the local label recommends permanent discontinuation) and exclusion criteria 10 (Evidence of any other disease, neurological or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of the investigational drug(s) or puts the patient at high risk for treatment-related complications).
- Anything else that is a major protocol deviation potentially impacting the primary endpoint (AE grade >=3 rates) or put patient at risk

#### 8.3 DEMOGRAPHIC AND BASELINE CHARACTERISTICS

The following information will be collected at screening examination ("baseline") between 14 days and 1 day before the first dose of study drug in this E-trial:

- Demographics: date of birth, gender, age in years, tumour type;
- P-trial information: P-trial protocol, dates of first and last dose of Bevacizumab, dose regimen on P-trial, other IMP treatments from P-trial.

All data for baseline characteristics and demographics will be listed. Patient characteristics (including indication) as well as demographics, will be summarized for the safety population by indication and overall.

### **8.4 MEDICAL HISTORY**

Medical History will not be coded. Only relevant medical history associated with a SAE is collected and will not be listed.

#### 8.5 PRIOR AND CONCOMITANT MEDICATION

Medications other than the study treatment will be recorded in the CRF if they are associated with a SAE and will not be listed.



Final version 3.0 / 18-FEB-2019

Concurrent P-trial anti-cancer IMP therapies will be referred as non-IMP treatment in this E-trial see section 8.6 for more details.

### 8.6 STUDY DRUG EXPOSURE AND/OR COMPLIANCE

#### 8.6.1 Bevacizumab Exposure

Treatment duration for Bevacizumab from E-trial will be estimated as follows:

Treatment Duration of Bevacizumab (E-trial) (months) = [(Date of last dose of Bevacizumab in E-trial – Date of first dose of Bevacizumab in E-trial) + 1] / 30.4375

Duration from first dose of Bevacizumab in P-trial to the last dose of Bevacizumab in the E-trial and derived approximate number of cycles of Bevacizumab will be also calculated. The derived approximate number of cycles of Bevacizumab will be calculated as the number of entire cycles, as follows:

Approximate number of cycles (overall) = [(Date of last dose of Bevacizumab in E-trial – Date of first dose of Bevacizumab in P-trial + 1) / (number of days in a cycle)],

where number of days in a cycle is the planned duration of cycle (14 or 21 days, depending of dose regimen).

Similarly, overall duration from first dose of Bevacizumab in P-trial to the last dose of Bevacizumab in the E-trial will be estimated as follows:

Treatment Duration of Bevacizumab (overall) (months) = [(Date of last dose of Bevacizumab in E-trial - Date of first dose of Bevacizumab in P-trial + 1) / 30.4375]

Duration of treatment of Bevacizumab (during E-trial and overall) and the derived number of cycles will be summarized for the safety population by indication and overall.

The dose received (mg/kg) and compliance will also be summarized for the E-trial full study duration (cumulative dose received). The summary will be presented overall and for each indication. To derive the dose received at a specific visit in mg/kg the dose received will be divided by the patient's weight (kg) at that visit, if the weight is missing it will be derived for the previous non-missing weight reported (i.e. last observation carried forward principle will be applied).

Cumulative dose of Bevacizumab = Sum (all doses of Bevacizumab within each cycle)

Compliance (%) = Dose received (mg/kg) / Planned Dose  $(mg/kg) \times 100$ .

The overall compliance will be derived using the cumulative dose received and the cumulative



Final version 3.0 / 18-FEB-2019

planned dose. The cumulative planned dose will not be adjusted for dose reduction or interruption (i.e. dose not administered).

Bevacizumab administration details with corresponding exposure will be presented in a listing. A flag will be presented in case the amount of dose is reduced for reasons other than a >10% change (loss or gain) in corresponding weight from baseline.

### 8.6.2 Non-IMP Exposure

Non-IMP administration details will be presented in a listing.

#### 8.7 EFFICACY DATA ENDPOINTS AND ANALYSES

The efficacy analysis will be performed on the safety population. No formal statistical testing is planned, so there will be no adjustment of the type I level for multiple endpoints.

All time to event efficacy endpoints defined in <u>section 8.7.1</u> and <u>section 8.7.2</u> will be calculated in days and converted to months considering the following conversion: 1 month = 30.4375 days.

### 8.7.1 Primary Efficacy Endpoint and Analyses

The primary variables will be based on the following safety endpoints: AE grade  $\geq$  3 related to Bevacizumab, SAEs and cause of death, Clopper-Pearson 95% CI will be derived for SAE incidence rates. Details on the summary of the primary endpoints are provided in section 8.10.1.

## 8.7.2 Secondary Efficacy Endpoints and Analysis

Assessments of efficacy will consist of assessments for progression of disease. Assessments for progression disease will be done as per the local standard, although it is recommended to continue using the same methods as in the P-trial. Results and dates of tumour assessments will be recorded. Assessment of progression of disease will be listed by indication, P-trial, country, center and patient.

### 8.7.2.1 Progression free survival

Progression free survival is defined as the time from first dose of Bevacizumab from E-trial to the time of first documented disease progression or death due to any cause, whichever occurs first. If a patient has not had an event, progression free survival is censored at the date of last tumour assessment. Time to event will be summarized in months (i.e. number of days/30.4375). The earliest date of disease progression will be used.

If a patient does not experience disease progression or did not die during the study then a censored progression free survival will be calculated as there will be no date of disease progression or date of death. This will be calculated as follows:



Final version 3.0 / 18-FEB-2019

Progression free survival (days) = (Date of last tumour assessment - Date of first dose of Bevacizumab from E-trial) + 1

If no tumour assessment is done for the patient the censoring day will be set to 1.

Progression free survival will be summarised using the Kaplan-Meier approach. The number of patients included in the analysis, with the event and without events (censored) as well as the minimum and maximum time to progression (including censored valued) will be summarized. Kaplan Meier estimates will be presented for:

- Median time to progression free survival, including 95% confidence Interval;
- 25% and 75% quartile;

In addition, a description of the survival rates in tabular form with the Kaplan Meier estimate of cumulative survival at relevant time points (eg 6, 12, 18, 24, 30 and >36 months) will also be presented. The final choice of the time points presented in the summary table might be updated dependent upon the data at the time of the analysis.

Finally, a graph with lines by indication of the Kaplan Meier survival function showing the event free probability, number of patients still at risk and censored observations.

The 95% confidence interval of the median estimate will be derived for each indication via the Greenwood method. The cumulative Kaplan Meier estimate will be presented at each time point, where the estimate will be from the closest, prior event (real or censored).

An exploratory analysis for progression free survival will be considered. For the exploratory analysis, progression free survival will be defined with reference to first dose of Bevacizumab from P-trial. Similar definitions and analysis will be considered as stated above for the corresponding progression free survival with reference to first dose of Bevacizumab from P-trial.

All progression free survival summaries and graphical representation will be performed by indication, if there are more than 5 patients in the indication.

#### 8.7.2.2 Overall survival time

Overall survival time is defined as the time from first dose of Bevacizumab from E-trial to death from any cause. Calculation is dependent on whether the patient dies or not and is measured in months i.e. (no. of days\*12)/365.25.

#### If a patient dies then:

Overall Survival Time = (Date of death – Date of first dose of Bevacizumab from E-trial) + 1



Final version 3.0 / 18-FEB-2019

**If a patient does not die during the study then** a censored overall survival time will be calculated as there will be no date of death. This will be calculated as follows:

Overall Survival Time = (Date of last known to be alive — Date of first dose of Bevacizumab in E-trial) + 1

Date of last known alive will be derived as the date of last contact if the patient is lost to follow-up or date of last visit if no safety follow-up was performed.

The same summaries as the ones provided for the progression free survival (see <u>section 8.7.2.1</u>), will be presented for the overall survival.

An exploratory analysis for overall survival will be considered. For the exploratory analysis, overall survival will be defined with reference to first dose of Bevacizumab from P-trial. Similar definitions and analysis will be considered as stated above for the corresponding overall survival with reference to first dose of Bevacizumab from P-trial.

All overall survival summaries and graphical representation will be performed by indication, if there are more than 5patients in the indication.

8.8 PHARMACOKINETIC/ PHARMACODYNAMIC ENDPOINTS AND ANALYSES

Not applicable.

8.9 QUALITY OF LIFE OR PHARMACOECONOMIC ENDPOINTS AND ANALYSES

Not applicable.

## 8.10 SAFETY DATA ENDPOINTS AND ANALYSES

#### 8.10.1 Adverse Events (AEs)

Adverse events recorded during the E-Trial (i.e. started after the first dose of Bevacizumab in the E-trial) will be summarized in frequency tables by primary system organ class and preferred term. All adverse events will be coded using the MedDRA dictionary. The version of the coding dictionary will be provided in the adverse events tables and listing footnote. Note: all AEs which started after the first dose of Bevacizumab in the E-trial are included in the AE summary and analyses tables.

The following adverse events are adverse events of special interest.

- Hypertension
- Reversible Posterior Leukoencephalopathy Syndrome (RPLS)



Final version 3.0 / 18-FEB-2019

- Proteinuria
- Haemorrhage, with a focus on haemoptysis and central nervous system (CNS) bleeding
- Arterial and venous thromboembolic events
- Wound healing complications
- Gastro-intestinal perforation
- Fistulae
- Congestive heart failure (CHF)

Roche will provide a complete list of preferred terms associated with each type of AE of special interest and will use this list to programmatically identify the AE's of special interest.

The number of patients, associated percentage and number of events will be presented for each indication, System Organ Class, Preferred Term, and overall.

- All adverse events
- AEs leading to discontinuation of Bevacizumab
- AEs leading to discontinuation of Bevacizumab/non-IMP
- Adverse events of special interest
- Adverse events leading to death
- Serious adverse events<sup>1</sup>
- Severe AEs related to Bevacizumab (grade 3-5)<sup>1</sup>

<sup>1</sup>95% confidence intervals of the incidence rate of the number of patients with at least one such AE is presented. The 95% confidence intervals will be based on Clopper-Pearson method.

The incidence rate shown in the adverse event tables will only be based on adverse events that started on or after the first treatment date in this E-trial.

A patient who experienced the same event on more than one occasion are counted only once in the calculation of counts of adverse events. Overall number of events will be counted in the event frequency.

For the incidence tables of adverse events related to Bevacizumab, adverse events leading to discontinuation of Bevacizumab, adverse events leading to discontinuation of Bevacizumab/non-IMP, adverse events of special interest, the frequency and percentage will be presented by maximum severity. For patients with more than one adverse event during the study of the same type, the maximum severity will be tabulated.

All adverse events will be listed by indication, P-trial, country, center and patient with the start and end date of the adverse event and corresponding study day, days since initial treatment date in P-trial, the severity and its relationship to the study treatment/non-IMP, action taken concomitant drug given and corresponding outcome. In addition, AEs of Special Interest and AEs ongoing from P-trials will be flagged on the listing.



Final version 3.0 / 18-FEB-2019

Separate listings will be provided for:

- All adverse events,
- Deaths

The number of patients who died, the cause of death, the relationship of death to Bevacizumab and relationship of death to non-IMP will be summarized overall and by P-trials.

**Laboratory Assessments** 

The laboratory results collected as part of the SAE report will be listed as recorded in the CRF. The pregnancy test results will also be listed.

### 8.10.2 Vital signs

Weight as a vital signs measurement will be assessed at baseline and prior to each cycle of Bevacizumab (and it will be collected only if dose of Bevacizumab was administered). Baseline body weight is used to calculate the starting dose in this E-trial. Baseline, for vital signs will be considered as the value measured at the cycle for which the first dose of Bevacizumab is administered.

### 8.10.3 Other safety data

Not applicable.

## 9 Interim Analyses

No formal interim analyses for efficacy is planned for this E-trial.

A formal interim safety analysis was done and reviewed from Medical perspective. Outputs can be made available upon request and are listed in Table 4.

## **10 Document History**

| Date | Version | Modified by | Brief details of changes made to template |
|---|---|---|---|
| 03-FEB-2015 | 1.0 | | Initial final version. |
| 20-SEP-2015 | 2.0 | | Added section after signature page (to match updated template) - The table of abbreviations for inclusion in the programmed outputs combined file. |
| | | | Section 6: specify that date imputation is only performed for AE and reason why, update name |



Final version 3.0 / 18-FEB-2019

| of the appendix to match appendix title. • Section 8.1 – update definition of follow-up time to be based on follow-up visit not disease progression (added censoring rules). Also added requirement to display 25% and 75% estimate of the follow-up time and number of patients with event/censored. Renamed to observation time. • Section 8.2 – Updated to include definition of a major protocol violation. • Sections 8.6.1 and 8.6.3.1 – Clarified in the derivations of exposure that the last dose date of |
|---|
| the non-IMP is not documented in the database |

• Section 8.10.1: clarify that only AE from the E-trial ((i.e. started after the first dose of Bevacizumab in the E-trial) are included in the summary tables. Added sentence to explain that all AE irrespective of start date compared to the last dose of treatment are included. Added that summary table of AEs ongoing from the P-trial, as well as a listing of AE related to non-IMP are required to interpret safety data.

date as the last dose of Bevacizumab.

and therefore this is assumed to be the same

- Section 8.10.3 updated the definition of baseline to match the first dose of Bevacizumab.
- Section 13.1:
  - Minor cosmetic update to the TFLs
  - o Footnote shortened to fit in one line.
  - Added Tables 1-1 to 3-1 for Roche publishing group (EudraCT format)
  - Post-text tables header added to all TFL to include date of data entry cut-off and date of data extraction
  - Post-text tables presenting data by indication and P-trial were split into 2 tables to help with the readability.
  - Tables 10-2 and 14.1.1-2 addition category for safety follow-up not performed added
  - Table 11-1 and 14.1.1-3 remove Tumor Type summary as included in the indication and remove the summary of duration of Bevacizumab in P trial and associated number of cycles are included in table 11-2 and 14.1.1-5.1.1.
  - O Added tables 14.3.1-1.9.1 and 14.3.1-1.9.2 as per update to section 8.10.1.
  - Added Listing 16.2-7.3 and renumbered subsequent listing.



Final version 3.0 / 18-FEB-2019

| 23-OCT-2015 | 2.1 | • Section 13.1: Minor cosmetic updates to following TFLs (Tables 14.1.1-5.2.1.1, 14.1.1-5.2.1.2, 14.1.1-5.1.1.1, 14.1.1-5.1.1.2, 14.1.1-2.1, 14.1.1-2.2, 14.1.1-5.2.3.1; Listing 16.2.5-1.2) |
|---|---|---|
| 21-JAN-2019 | 2.2 | SAP text and TFL shells revised for upcoming final analysis. |
| 18-FEB-2019 | 3.0 | Finalized v3.0 of SAP. |

## 11 References

None

# **12 Appendices**

12.1 Tables, Figures and Listing shells



**Statistical Analysis Plan:** Final version 3.0 / 18-FEB-2019

**Table 4.** List of Tables, Figures and Listings for the Clinical Study Report

| Output<br>Type | Number | Title | Included in IA? |
|---|---|---|---|
| IN-TEXT | | | |
| Table | <u>10-1</u> | P-trials Contribution to the E-trial | N |
| Table | <u>10-2</u> | Patient Disposition | N |
| Table | <u>11-1</u> | Demographics and Baseline Characteristics | N |
| Table | <u>11-2</u> | Duration and Exposure to Bevacizumab | γ* |
| Table | <u>11-3</u> | Bevacizumab Overall Compliance | N |
| Table | <u>12-1</u> | Number (%) of Patients with Adverse Events by System Organ Class and Preferred Term (Incidence ≥ 5% in any Indication) | N |
| Table | <u>12-2</u> | Number (%) of Patients with Adverse Events of Special Interest (AESI) by AESI Category and Preferred Term | N |
| Table | <u>12-3</u> | Cause of Death and Relationship of Death to Study Treatment | N |
| Table | <u>1-1</u> | Demographics by Indication (EudraCT Format) | N |
| Table | <u>2-1</u> | Serious Adverse Events by Indication (EudraCT Format) | N |
| Table | <u>3-1</u> | Non-Serious Adverse Events reported in >=5% of subjects in any indication by Indication (EudraCT Format) | N |
| POST-TE | хт | | |
| Section 1 | 14.1 Demographic | cs and Baseline Characteristics | |
| Table | <u>14.1.1-1</u> | P-trials Contribution to the E-trial (All Patients Population) | Υ |
| Table | 14.1.1-2.1 | Patient Disposition by Indication (All Patients Population) | Y |
| Table | 14.1.1-3.1 | Demographics and Baseline Characteristics by Indication (All Patients Population) | Y |
| Table | 14.1.1-4.1 | Major Protocol Deviations by Indication (All Patients Population) | N |
| Table | 14.1.1-5.1.1.1 | Duration and Exposure to Bevacizumab by Indication (Safety Population) | Υ* |
| Table | 14.1.1-5.1.2.1 | Bevacizumab Compliance by Indication (Safety Population) | N |
| Section 1 | 14.2 Efficacy | | · |
| Table | <u>14.2-1.1</u> | Progression Free Survival (PFS) by Indication (Safety Population) | N |

 BMSOP111/F2



**Statistical Analysis Plan:** Final version 3.0 / 18-FEB-2019

| Output<br>Type | Number | Title | Included in IA? |
|---|---|---|---|
| Table | <u>14.2-1.2</u> | Overall Survival (OS) by Indication (Safety Population) | N |
| Table | 14.2-1.3 | Progression Free Survival (PFS) by Indication - Exploratory analysis, PFS with reference to first dose of Bevacizumab from P-trial (Safety Population) | N |
| Table | 14.2-1.4 | Overall Survival (OS) by Indication - Exploratory analysis, OS with reference to first dose of Bevacizumab from P-trial (Safety Population) | N |
| Figure | <u>14.2-1.1</u> | Progression Free Survival (PFS) by Indication (Safety Population) | N |
| Figure | <u>14.2-1.2</u> | Overall Survival (OS) by Indication (Safety Population) | N |
| Figure | <u>14.2-1.3</u> | Progression Free Survival (PFS) by Indication - Exploratory analysis, PFS with reference to first dose of Bevacizumab from P-trial (Safety Population) | N |
| Figure | 14.2-1.4 | Overall Survival (OS) by Indication - Exploratory analysis, OS with reference to first dose of Bevacizumab from P-trial (Safety Population) | N |
| Section 1 | L4.3 Safety | | |
| Section 1 | L4.3.1 Adverse Ev | vents | |
| Table | 14.3.1-1.1.1 | Number (%) of Patients with Adverse Events by Indication, System Organ Class and Preferred Term (Safety Population) | Υ |
| Table | 14.3.1-1.1.2 | Number (%) of Patients with Severe (Grade 3-5) Adverse Events Related to Bevacizumab by Indication, System Organ Class and Preferred Term (Safety Population) | |
| Table | 14.3.1-1.2.1 | Number (%) of Patients with Adverse Events Related to Bevacizumab by Indication, System Organ Class, Preferred Term and Maximum Severity (Safety Population) | Υ |
| Table | 14.3.1-1.3.1 | Number (%) of Patients with Adverse Events Leading to Discontinuation of Bevacizumab by Indication, System Organ Class and Preferred Term (Safety Population) | N |
| Table | 14.3.1-1.3.2 | Number (%) of Patients with Adverse Events Leading to Discontinuation of Bevacizumab/non-IMP by Indication, System Organ Class and Preferred Term (Safety Population) | N |
| Table | 14.3.1-1.4.1 | Number (%) of Patients with Adverse Events Leading to Discontinuation of Bevacizumab by Indication, System Organ Class, Preferred Term and Maximum Severity (Safety Population) | N |
| Table | 14.3.1-1.4.2 | Number (%) of Patients with Adverse Events Leading to Discontinuation of Bevacizumab/non-IMP by Indication, System Organ Class, Preferred Term and Maximum Severity (Safety Population) | N |
| Table | 14.3.1-1.5.1 | Number (%) of Patients with Adverse Events of Special Interest (AESI) by Indication, AESI Category and Preferred Term (Safety Population) | Υ |
| Table | 14.3.1-1.6.1 | Number (%) of Patients with Adverse Events of Special Interest (AESI) by Indication, AESI Category, Preferred Term and Maximum Severity (Safety Population) | Y |

 BMSOP111/F2



**Statistical Analysis Plan:** Final version 3.0 / 18-FEB-2019

| Output<br>Type | Number | Title | Included in IA? |
|---|---|---|---|
| Table | 14.3.1-1.7.1 | Number of Adverse Events Leading to Death by Indication, System Organ Class, Preferred Term and Outcome (Safety Population) | γ* |
| Table | 14.3.1-1.8.1 | Number (%) of Patients with Non-Serious Adverse Events by Indication, System Organ Class, Preferred Term (Incidence ≥ 5% in any Indication) (Safety Population) | |
| Table | 14.3.1-2.1 | Number (%) of Patients with Serious Adverse Events by Indication, System Organ Class and Preferred Term (Safety Population) | Υ |
| Table | 14.3.1-2.2 | Number (%) of Patients with Severe (Grade 3-5) Adverse Events Related to Bevacizumab by Indication, System Organ Class and Preferred Term (Safety Population) | γ* |
| Table | 14.3.1-4.1 | Cause of Death and Relationship of Death to Study Treatment by Indication (Safety Population) | Y |
| Section 1 | 6.2 Listings | | |
| Section 1 | .6.2.1 End of Stu | dy | |
| Listing | <u>16.2.1-1</u> | End of Treatment/Study (All Patients Population) | γ* |
| Section 1 | .6.2.2 Protocol D | eviations | |
| Listing | <u>16.2.2-1</u> | Protocol Deviations (All Patients Population) | N |
| Section 1 | .6.2.3 Analysis Po | ppulations | |
| Section 1 | .6.2.4 Demograp | hics and Baseline Characteristics | |
| Listing | <u>16.2.4-1.1</u> | Demographics and Baseline Characteristics (All Patients Population) | Υ |
| Listing | 16.2.4-1.2 | P-trial Information (All Patients Population) | γ* |
| Listing | 16.2.4-2 | Pregnancy Test (All Patients Population) | N |
| Section 1 | 6.2.5 Study Drug | g Administration | |
| Listing | 16.2.5-1.1 | Administration of Bevacizumab (Safety Population) | γ* |
| Listing | 16.2.5-1.2 | Administration of non-IMP Treatment (Safety Population) | Υ |
| Listing | <u>16.2.5-2</u> | Duration of exposure to Bevacizumab (Safety Population) | N |
| Section 1 | 6.2.6 Efficacy | | |
| Listing | 16.2.6-1.1 | Time to Event (Safety Population) | N |
| Listing | 16.2.6-1.2 | Progression Assessment (Safety Population) | N |
| Section 1 | 6.2.7 Adverse Ev | vents | |


 BMSOP111/F2



Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

| Output<br>Type | Number | Title | Included in IA? |
|---|---|---|---|
| Listing | <u>16.2.7-1</u> | Adverse Events (Safety Population) | γ* |
| Listing | 16.2.7-2 | All Deaths (Safety Population) | γ* |

Included in IA: N=No; Y=Yes; Y\*=Yes, however shell was updated in version 3.0 of the SAP.

To note further TFLs were presented in the IA, as documented in version 2.0 of the SAP. For final analysis, all TFLs defined in final version 3.0 of the SAP will be presented.



**Statistical Analysis Plan:** Final version 3.0 / 18-FEB-2019

## 12.1.1 In-text Tables, Figures and Listing shells

**Table 10-1 P-trials Contribution to the E-trial** 

| P-Trials | ВС | OC or PC | CRC | RCC | NSCLC | GBM | Total |
|---|---|---|---|---|---|---|---|
| Any P-trials | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| xxxxxx | XX (XX.X%) | | | | | | XX (XX.X%) |
| XXXXXX | , | | | XX (XX.X%) | | | XX (XX.X%) |
| XXXXXX | | XX (XX.X%) | | , , | XX (XX.X%) | | XX (XX.X%) |
| XXXXXX | | XX (XX.X%) | | | , | XX (XX.X%) | XX (XX.X%) |
| XXXXXX | | , , | XX (XX.X%) | | | , | XX (XX.X%) |
| XXXXXX | | | XX (XX.X%) | | | | XX (XX.X%) |
| XXXXXX | | | XX (XX.X%) | | | | XX (XX.X%) |
| XXXXXX | XX (XX.X%) | | , | | | | XX (XX.X%) |
| (cont.) | , , | | | | | | XX (XX.X%) |

Source: Table 14.1.1-1



**Table 10-2 Patient Disposition** 

Final version 3.0 / 18-FEB-2019

| | BC<br>(N=XX) | OC or PC<br>(N=XX) | CRC<br>(N=XX) | RCC<br>(N=XX) | NSCLC<br>(N=XX) | GBM<br>(N=XX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|---|
| Enrolled | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Treated (Safety Population) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| ` • • • • | XX (XX.X%) | XX (XX.X%) | ` , | XX (XX.X%) | XX (XX.X%) | ` , | , |
| Ongoing<br>Discontinued | , | | XX (XX.X%) | , | ` , | XX (XX.X%) | XX (XX.X%) |
| | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| SFU visit performed | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| SFU visit not perfromed | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Reason for discontinuation fro | m Bevacizumab tr | eatment: | | | | | |
| Adverse event | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Disease progression | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Withdrawal of consent | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Death | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Lack of compliance | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X% |
| (cont.) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Reason follow-up not complet | ed· | | | | | | |
| Withdrawal of consent | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Lost to follow-up | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Death | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| (cont.) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| (COTIL.) | XX (XX.X70) | XX (XX.X70) | XX (XX.X70) | XX (XX.X70) | XX (XX.X70) | XX (XX.X70) | XX (XX.X70) |
| Observation Time (Months)* | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| (95% CI) | (XX.X; XX.X) | (XX.X; XX.X) | (XX.X; XX.X) | (XX.X; XX.X) | (XX.X; XX.X) | (XX.X; XX.X) | (XX.X; XX.X |
| (25%; 75%) | (XX.X; XX.X) | (XX.X; XX.X) | (XX.X; XX.X) | (XX.X; XX.X) | (XX.X; XX.X) | (XX.X; XX.X) | (XX.X; XX.X |

<sup>\*</sup> Onbervation time is defined as time to safety follow-up – first bev. admin in E-trial based on inverse KM. Abbreviations: KM=Kaplan-Meier; SFU=Safety Follow-up; SE=Standard error.

Source: Table 14.1.1-2.1




Final version 3.0 / 18-FEB-2019

**Table 11-1 Demographics and Baseline Characteristics** 

| | BC<br>(N=XXX) | OC or PC<br>(N=XXX) | CRC<br>(N=XXX) | RCC<br>(N=XXX) | NSCLC<br>(N=XXX) | GBM<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|---|
| Gender | | | | | | | |
| Female | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Male | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Age (years) | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X ` | XX.X ` | XX.X ` | XX.X ` | XX.X ` | XX.X ` | XX.X ` |
| [Min; Max] | [XX; XX] | [XX; XX] | [XX; XX] | [XX; XX] | [XX; XX] | [XX; XX] | [XX; XX] |
| Veight at baseline (kg) | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X ` | XX.X ` | XX.X ` | XX.X ` | XX.X ` | XX.X ` | XX.X ` |
| [Min; Max] | [XX; XX] | [XX; XX] | [XX; XX] | [XX; XX] | [XX; XX] | [XX; XX] | [XX; XX] |

Source: Table 14.1.1-3.1



Final version 3.0 / 18-FEB-2019

**Table 11-2 Duration and Exposure to Bevacizumab** 

| | BC<br>(N=XXX) | OC or PC<br>(N=XXX) | CRC<br>(N=XXX) | RCC<br>(N=XXX) | NSCLC<br>(N=XXX) | GBM<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|---|
| Treatment Duration of Bev | acizumab (E-trial) * (Month: | s) | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| [Min; Max] | [XX.X; XX.X] | [XX.X; XX.X]<br>XX | [XX.X; XX.X]<br>XX | [XX.X; XX.X]<br>XX | [XX.X; XX.X]<br>XX | [XX.X; XX.X]<br>XX | [XX.X; XX.X]<br>XX |
| Treatment Duration of Bev | acizumab (overall) ** (Mont | hs) | | | | | |
| n | XX ´ ` | ΧX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) |
| Median | XX.XX ` | XX.XX ` | XX.XX ` | XX.XX ` | XX.XX ` | XX.XX ` | XX.XX ` |
| [Min; Max] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] |
| Approximate number of cy | cles (overall) *** [n (%)] | | | | | | |
| 1-10 | ` XX (XX.X%)´ | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 11-20 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 21-30 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 31-40 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 41-50 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 51-60 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| (cont.) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

#### Note

Source: Table 14.1.1-5.1.1.1


BMSOP111/F2

<sup>\*</sup> Treatment Duration of Bev. (E-trial) = [(Date of last dose of Bev. in E-trial - Date of first dose of Bev. in E-trial) + 1]/30.4375.

<sup>\*\*</sup> Treatment Duration of Bev. (overall) = [(Date of last dose of Bev. in E-trial – Date of first dose of Bev. in P-trial) + 1]/30.4375.

<sup>\*\*\*</sup> Approximate number of cycles (overall) = [(Date of last dose of Bev. in E-trial – Date of first dose of Bev. in P-trial) + 1] / (number of days in a cycle).



Final version 3.0 / 18-FEB-2019

**Table 11-3 Bevacizumab Overall Compliance** 

| | BC<br>(N=XXX) | OC or PC<br>(N=XXX) | CRC<br>(N=XXX) | RCC<br>(N=XXX) | NSCLC<br>(N=XXX) | GBM<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|---|
| Dose Received (mg/kg) | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X ` | XX.X ` | XX.X ` | XX.X ` | XX.X` | XX.X` | XX.X` |
| [Min; Max] | [XX; XX] | [XX; XX] | [XX; XX] | [XX; XX] | [XX; XX] | [XX; XX] | [XX; XX] |
| Compliance (%) | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X ` | XX.X ` | XX.X ` | XX.X ` | XX.X ` | XX.X` | XX.X ` |
| [Min; Max] | [XX; XX] | [XX; XX] | [XX; XX] | [XX; XX] | [XX; XX] | [XX; XX] | [XX; XX] |
| Compliance [n (%)] | | | | | | | |
| < 80% | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| 80 - 120% | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| > 120% | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | , | , , | ` , | , | , | , | ` , |

Source: Table 14.1.1-5.1.2.1



Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

Table 12-1 Number (%) of Patients with Adverse Events by System Organ Class and Preferred Term (Incidence ≥ 5% in any Indication)

| System Organ Class/<br>Preferred Term | BC<br>(N=XX)<br>n (%) [Events] | OC or PC<br>(N=XX)<br>n (%) [Events] | CRC<br>(N=XX)<br>n (%) [Events] | RCC<br>(N=XX)<br>n (%) [Events] | NXCLC<br>(N=XX)<br>n (%) [Events] |
|---|---|---|---|---|---|
| Any System Organ Class | XX (XXX.X) [XXX] | XX (XXX.X) [XXX] | XX (XXX.X) [XXX] | XX (XXX.X) [XXX] | XX (XXX.X) [XXX] |
| System Organ Class 1 | XX (XXX.X) [XXX] | XX (XXX.X) [XXX] | XX (XXX.X) [XXX] | XX (XXX.X) [XXX] | XX (XXX.X) [XXX] |
| Preferred Term 1 | XX (XXXXX) [XXX] | XX (XXXXX) XXX | XX (XXX.X) [XXX] | XX (XXX.X) [XXX] | XX (XXXX) [XXX] |
| Preferred Term 2 | [XXX] (X.XXX) XX | XX (XXXXX) [XXX] | XX (XXX.X) [XXX] | XX (XXXXX) [XXX] | XX (XXX.X) [XXX] |
| Preferred Term 3 | [XXX] (X.XXX) XX | XX (XXX.X) [XXX] | XX (XXX.X) [XXX] | XX (XXX.X) [XXX] | XX (XXX.X) [XXX] |
| (cont.) | xx (xxxxx) [xxx] | xx (xxx.x) [xxx] | xx (xxx.x) [xxx] | xx (xxx.x) [xxx] | xx (xxx.x) [xxx] |
| (cont.) | XX (XXX.X) [XXX] | XX (XXX.X) [XXX] | XX (XXX.X) [XXX] | XX (XXX.X) [XXX] | XX (XXX.X) [XXX] |

Note:

MedDRA version <

A patient with multiple occurrences of an AE is counted only once in each SOC and/or PT.

Source: Table 14.3.1-1.1.1

#### Programming Note:

- Include all Indications (additional columns), including Total - If possible fit all in one page.

Template Author: Version 3.0 16AUG2017  BMSOP111/F2



Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

Table 12-2 Number (%) of Patients with Adverse Events of Special Interest (AESI) by AESI Category and Preferred Term

| AESI Category/<br>Preferred Term | BC<br>(N=XX)<br>n (%) [Events] | OC or PC<br>(N=XX)<br>n (%) [Events] | CRC<br>(N=XX)<br>n (%) [Events] | RCC<br>(N=XX)<br>n (%) [Events] | NXCLC<br>(N=XX)<br>n (%) [Events] |
|---|---|---|---|---|---|
| Any AESI | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] |
| Hypertension | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] |
| Preferred Term 1 | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX |
| Preferred Term 2 | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] |
| Preferred Term 3 | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX |
| (cont.) | xx (xxx.x) [xx] | xx (xxx.x) [xx] | xx (xxx.x) [xx] | xx (xxx.x) [xx] | xx (xxx.x) [xx] |
| (cont.) | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] |

Note:

MedDRA version <

A patient with multiple occurrences of an AE is counted only once in each AESI category and/or PT. A PT can contribute to more than one AESI category.

Source: Table 14.3.1-1.5.1

#### Programming Note:

- Include all Indications (additional columns), including Total




**Statistical Analysis Plan:** Final version 3.0 / 18-FEB-2019

Table 12-3 Cause of Death and Relationship of Death to Study Treatment

| | BC<br>(N=XXX) | OC or PC<br>(N=XXX) | CRC<br>(N=XXX) | RCC<br>(N=XXX) | NSCLC<br>(N=XXX) | GBM<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|---|
| No of patients who died | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Cause of death* | | | | | | | |
| Progressive disease | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Adverse event | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Other | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Relationship of death to Bevacizumab* | | | | | | | |
| Related | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Unrelated | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Relationship of death to Other Non-IMP* | | | | | | | |
| Related | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |
| Unrelated | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) | XXX (XX.X%) |

<sup>\*</sup> Percentages are calculated from the number of patients who died within the indication considered.

Source: Table 14.3.1-4.1




Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

### 12.1.2 EudraCT Tables

Table 1-1 Demographics by Indication (EudraCT Format) (All Patients population)

| | BC<br>(N=XXX)<br>n (%) | OC or PC<br>(N=XXX)<br>n (%) | CRC<br>(N=XXX)<br>n (%) | RCC<br>(N=XXX)<br>n (%) | NSCLC<br>(N=XXX)<br>n (%) | GBM<br>(N=XXX)<br>n (%) | Total<br>(N=XXX)<br>n (%) |
|---|---|---|---|---|---|---|---|
| Age | | | | | | | |
| 18-64 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 65-84 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| 85+ | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Total | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Country | | | | | | | |
| Country #1 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Country #2 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Country #3 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| (cont.) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Total | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |

Source: Listing 16.2.4-1.1

Program Name: xxxxxxx Page X of Y


 BMSOP111/F2


Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

Table 2-1 Serious Adverse Events by Indication (EudraCT Format) (Safety Population)

| System Organ Class | BC<br>(N=XXX) | | | | | | | OC or P | | | CRC<br>(N=XXX) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Preferred Term | NSUB | NEVS | NTRE | NERD | NTRD | NSUB | NEVS | NTRE | NERD | NTRD | NSUB | NEVS | NTRE | NERD | NTRD |
| Number of subjects with at least one serious adverse | ı | | | | | | | | | | | | | | |
| event | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| SOC 1 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| PT 1 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| PT 2 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| SOC 2 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| PT 1 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| PT 2 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| 2000 | | | | | | | | | | | | | | | |

NSUB=Number of Subjects with Event, NEVS=Number of Events, NTRE=Number of Treatment Related Events, NERD=Number of Events Resulting in Death, NTRD=Number of Treatment Related Events Resulting in Death

Source: Listing XXXX

Program Name: xxxxxxxx Page X of Y

# Programming Note:

- Repeat for all indication + total
- Sort by decreasing frequency for SOC and PT.




Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

Table 3-1 Non-Serious Adverse Events reported in >=5% of subjects in any indication by Indication (EudraCT Format) (Safety population)

| | (N | BC<br>=XXX) | | or PC<br>=XXX) | | CRC<br>(N=XXX) |
|---|---|---|---|---|---|---|
| System Organ Class Preferred Term | Number (%)<br>of Subjects | Number of events | Number (%) of<br>Subjects | Number of events | Number (%) of<br>Subjects | Number of events |
| Number of subjects with at least one non-serious adverse events reported in >=5% of subjects | XXX (XX.X) | XXX | XXX (XX.X) | XXX | XXX (XX.X) | XXX |
| SOC 1 | XXX (XX.X) | XXX | XXX (XX.X) | XXX | XXX (XX.X) | XXX |
| PT 1 | XXX (XX.X) | XXX | XXX (XX.X) | XXX | XXX (XX.X) | XXX |
| PT 2 | XXX (XX.X) | XXX | XXX (XX.X) | XXX | XXX (XX.X) | XXX |
| GARAGE CONTRACTOR CONT | XXX (XX.X) | XXX | XXX (XX.X) | XXX | XXX (XX.X) | XXX |
| SOC 2 | XXX (XX.X) | XXX | XXX (XX.X) | XXX | XXX (XX.X) | XXX |
| PT 1 | XXX (XX.X) | XXX | XXX (XX.X) | XXX | XXX (XX.X) | XXX |
| PT 2 | XXX (XX.X) | XXX | XXX (XX.X) | XXX | XXX (XX.X) | XXX |
| | XXX (XX.X) | XXX | XXX (XX.X) | XXX | XXX (XX.X) | XXX |

Source: Listing XXXXX

Program Name: xxxxxxx Page X of Y

#### Programming Note:

- Repeat for all indications + total
- Sort by decreasing frequency for SOC and PT.
- MUST EXCLUDE any SAEs
- Organized by SOC, then preferred term that occurred at a frequency of >= 5% for the indication considered. The table should also include the following:
  - o Total number of patients with at least 1 non-serious AE (per indication applying the >= 5% threshold; i.e., reflective of ONLY the terms included in the table)
  - o Number of patients with each non-serious AE (at the >= 5% threshold) by treatment group
- Number of EVENTS for each preferred term by treatment group

Template Author:
Version 3.0 16AUG2017

 BMSOP111/F2



Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

# 12.1.3 Post-text Tables, Figures and Listing shells

M025757 -- DELIVERY TYPE -- Page X of Y

Table 14.1.1-1
P-trials Contribution to the E-trial
(All Patients Population)

| P-Trial/<br>Center | BC<br>(N=XX)<br>n (%) | OC or PC<br>(N=XX)<br>n (%) | CRC<br>(N=XX)<br>n (%) | RCC<br>(N=XX)<br>n (%) | NSCLC<br>(N=XX)<br>n (%) | GBM<br>(N=XX)<br>n (%) | Total<br>(N=XX)<br>n (%) |
|---|---|---|---|---|---|---|---|
| Any P-trial | xx (xxx.x) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| AVF3694g | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| XXXXX | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| XXXXX | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| XXXXX<br>(cont.) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| XXXXXX | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| XXXXX | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| XXXXX | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| XXXXX (cont.) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |

Note: Percentages at a center level are based on the number of patients enrolled from the corresponding P-trial.

Source : Listing XXXXXX

<Program Path\Program name.sas> <run on: datetime>

# Programming Note:

Include all P-trials.




Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

Page X of Y

M025757 -- DELIVERY TYPE -- Table 14.1.1-2.1

Patient Disposition by Indication (All Patients Population)

| | BC | OC or PC | CRC | RCC | NSCLC |
|---|---|---|---|---|---|
| | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Enrolled [n (%)] | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Preated (Safety Population) [n (%)] | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Ongoing [n(%)] | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Discontinued [n(%)] | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| SFU visit performed [n(%)] | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| SFU visit not performed [n(%)] | | | | | |
| Reason for discontinuation from Bevacizuma | o treatment: [n(%)] | | | | |
| Adverse event | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| (cont.) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Reason follow-up not completed: [n(%)] | | | | | |
| Withdrawal of consent | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Death | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| (cont.) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Other | | | | | |
| Observation Time (Months)* | | | | | |
| n | XX | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| (95% CI) | (XX.X; XX.X) | (XX.X; XX.X) | (XX.X; XX.X) | (XX.X; XX.X) | (XX.X; XX. |
| (25%; 75%) quartiles | (XX.X; XX.X) | (XX.X; XX.X) | (XX.X; XX.X) | (XX.X; XX.X) | (XX.X; XX. |

Note: \* Observation time is defined as time to safety follow-up - first bev. admin in E-trial based on inverse KM. Abbreviations: KM=Kaplan-Meier; SFU=Safety Follow-up; SE=Standard error.

Source : Listing XXXXXX

<Program Path\Program name.sas> <run on: datetime>

# Programming Note:

- Include all Indications (additional columns), including Total, if possible try to fit all column in 1 page
- List only the reasons for discontinuation that are populated.




Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

Page 1 of Y

M025757 -- DELIVERY TYPE -- Table 14.1.1-3.1

Table 14.1.1-3.1

Demographics and Baseline Characteristics by Indication (All Patients Population)

| | BC<br>(N=XX) | OC or PC (N=XX) | CRC (N=XX) | RCC (N=XX) | NSCLC<br>(N=XX) |
|---|---|---|---|---|---|
| Gender [n (%)] | | | | | |
| Female | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Male | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Age (years) | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| [Min; Max] | [XX; XX] | [XX; XX] | [XX; XX] | [XX; XX] | [XX; XX] |
| Weight at baseline (kg) | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| [Min; Max] | [XX; XX] | [XX; XX] | [XX; XX] | [XX; XX] | [XX; XX] |

Source : Listing XXXXXX

<Program Path\Program name.sas> <run on: datetime>

# Programming Note:

- Include all Indications (additional columns), including Total, if possible try to fit all column in 1 page
- Display summary statistics with 0 dp for weight and 0 dp for age.




Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

Page X of Y

M025757 -- DELIVERY TYPE -- Table 14.1.1-4.1

Major Protocol Deviations by Indication (All Patients Population)

| | BC<br>(N=XX)<br>n (%) | | OC or PC<br>(N=XX)<br>n (%) | | (N= | =XX) | RCC<br>(N= | =XX) | NSC<br>(N=<br>n | XX) |
|---|---|---|---|---|---|---|---|---|---|---|
| | | ( - / | 2.55 | | | () | | ( - / | ==/. 0 | |
| Any major protocol deviations | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) |
| Inclusion criteria | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) |
| Protocol Deviation 2 | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) |
| Protocol Deviation 3 | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) |
| Exclusion Criteria | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) |
| Protocol Deviation 8 | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) |
| Protocol Deviation 10 | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) |
| Not compliant to Bevacizumab treatment | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) |
| Not allowed medications | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) |
| (cont.) | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) | XX | (XXX.X) |

Source : Listing XXXXXX

<Program Path\Program name.sas> <run on: datetime>

# Programming Note:

- Include all Indications (additional columns), including Total, if possible try to fit all column in 1 page
- Included in summary major protocol deviations from :
  - o inclusion criteria 2 (Patient is treated with bevacizumab at the end of the Roche/Genentech sponsored P-trial and continues to have benefit as judged by the investigator) and inclusion criteria 3 (Eligible for continuation of bevacizumab treatment at the end of the P-trial, according to P-trial protocol);
  - o exclusion criteria 8 (Evidence of any AE potentially attributable to bevacizumab, for which the local label recommends permanent discontinuation) and exclusion criteria 10 (Evidence of any other disease, neurological or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of the investigational drug(s) or puts the patient at high risk for treatment-related complications)


 BMSOP111/F2



Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

o anything else that is a major protocol deviation potentially impacting the primary endpoint (AE grade >=3 rates) or put patient at risk.




**Statistical Analysis Plan:** Final version 3.0 / 18-FEB-2019

Page X of Y

M025757 -- DELIVERY TYPE -- Table 14.1.1-5.1.1.1

Duration and Exposure to Bevacizumab by Indication (Safety Population)

| | BC | OC or PC | CRC | RCC | NSCLC |
|---|---|---|---|---|---|
| | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Treatment Duration of Bevac | cizumab (E-trial) * (Months) | | | | |
| n | XX.X | XX.X | XX.X | XX.X | XX.X |
| Mean (SD) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| [Min; Max] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] |
| Treatment Duration of Bevac | cizumab (overall) ** (Months) | | | | |
| n | XX.X | XX.X | XX.X | XX.X | XX.X |
| Mean (SD) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| [Min; Max] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] |
| Approximate number of cycle | es (overall) *** [n (%)] | | | | |
| 1-10 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| 11-20 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| 21-30 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| 31-40 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| 41-50 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| 51-60 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| (cont.) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |

Note: \* Treatment Duration of Bev. (E-trial) = [(Date of last dose of Bev. in E-trial - Date of first dose of Bev. in E-trial) + 1]/30.4375.

Source : Listing XXXXXX

<Program Path\Program name.sas> <run on: datetime>


 BMSOP111/F2

<sup>\*\*</sup> Treatment Duration of Bev. (overall) = [(Date of last dose of Bev. in E-trial - Date of first dose of Bev. in P-trial) + 1]/30.4375.

<sup>\*\*\*</sup> Approximate number of cycles (overall) = [(Date of last dose of Bev. in E-trial - Date of first dose of Bev. in P-trial) + 1] / (number of days in a cycle).



Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

# Programming Note:

- Include all Indications (additional columns), including Total, if possible try to fit all column in 1 page.
- Display treatment duration with 1dp.




Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

Page X of Y

M025757

# -- DELIVERY TYPE -Table 14.1.1-5.1.2.1 Bevacizumab Compliance by Indication (Safety Population)

| | BC | | CRC | RCC | NSCLC |
|---|---|---|---|---|---|
| | (N=XX) | OC or PC (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Dose Received (mg/kg) | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| [Min; Max] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] |
| Compliance (%) | | | | | |
| n | XX | XX | XX | XX | XX |
| Mean (SD) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) | XX.XX (XX.XXX) |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| [Min; Max] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] | [XX.X; XX.X] |
| Compliance [n (%)] | | | | | |
| < 80% | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| 80 - 120% | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| > 120% | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |

Source : Listing XXXXXX

<Program Path\Program name.sas> <run on: datetime>

# Programming Note:

- Include all Indications (additional columns), including Total, if possible try to fit all column in 1 page
- Repeat for all cycles.

 BMSOP111/F2



Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

Page X of Y

M025757 -- DELIVERY TYPE -- Table 14.2-1.1

Progression Free Survival (PFS) by Indication (Safety Population)

Indication: XXXXX

| | Bevacizumab<br>Total<br>(N=XX) |
|---|---|
| Number of patients [n (%)] [a] | |
| who were censored | XXX (XXX.X) |
| who did have disease progression or died | XXX (XXX.X) |
| Time to disease progression (months) [b] | |
| Mean (SD) | XX.XX (XX.XXX) |
| Q1 | XX.X |
| Median (95% CI) | XX.X (XX.X, XX.X) |
| Q3 | XX.X |
| [Min; Max] | [XX.X; XX.X] |
| Estimated probabilities of progression (95% CI) [c] | |
| 6 months | XX (XX.X, XX.X) |
| 12 months | XX (XX.X, XX.X) |
| (cont.) | |

- [a] Percentages are based on the number of patients in the Safety population.
- [b] Estimates are from a Kaplan-Meier analysis.
- [c] 95% CI (confidence interval) for the estimated probability are derived using Greenwood method.

PFS calculated with reference to first dose of Bevacizumab from E-trial.

Source : Listing XXXXXX

<Program Path\Program name.sas> <run on: datetime>

# Programming Note:

- Repeat for all indications, if > 5 patients are included in the considered indication.




Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

Page X of Y

M025757 -- DELIVERY TYPE -Table 14.2-1.2
Overall Survival (OS) by Indication
(Safety Population)

Indication: XXXXX

| | Bevacizumab<br>Total<br>(N=XX) |
|---|---|
| Number of patients [n (%)] [a] | |
| who were censored | XXX (XXX.X) |
| who died | XXX (XXX.X) |
| Time to death (months) [b] | |
| Mean (SD) | XX.XX (XX.XXX) |
| Q1 | XX.X |
| Median (95% CI) | XX.X (XX.X, XX.X) |
| Q3 | XX.X |
| [Min; Max] | [XX.X; XX.X] |
| Estimated probabilities of death (95% CI) [c] | |
| 6 months | XX (XX.X, XX.X) |
| 12 months | XX (XX.X, XX.X) |
| (cont.) | |

- [a] Percentages are based on the number of patients in the Safety population.
- [b] Estimates are from a Kaplan-Meier analysis.
- [c] 95% CI (confidence interval) for the estimated probability are derived using Greenwood method.
- OS calculated with reference to first dose of Bevacizumab from E-trial.

Source : Listing XXXXXX

<Program Path\Program name.sas> <run on: datetime>

# Programming Note:

- Repeat for all indications, if > 5 patients are included in the considered indication.




Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

Table 14.2-1.3

Progression Free Survival (PFS) by Indication - Exploratory analysis, PFS with reference to first dose of Bevacizumab from P-trial (Safety Population)

# Programming Note:

- Replicate of Table 14.2-1.1.
- Updated last footnote to the following: PFS calculated with reference to first dose of Bevacizumab from P-trial.

Table 14.2-1.4

Overall Survival (OS) by Indication - Exploratory analysis, OS with reference to first dose of Bevacizumab from P-trial (Safety Population)

# Programming Note:

- Replicate of Table 14.2-1.2.
- Updated last footnote to the following: OS calculated with reference to first dose of Bevacizumab from P-trial.

 BMSOP111/F2



Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

Page X of Y

M025757 -- DELIVERY TYPE -- Figure 14.2-1.1

Progression Free Survival (PFS) by Indication (Safety Population)



PFS calculated with reference to first dose of Bevacizumab from E-trial.

Source : Listing XXXXXX

<Program Path\Program name.sas> <run on: datetime>

# Programming Note:

- X-axis Label "Progression free survival (Months)"
- Y-axix Label "Survival probability (%).
- Present "Median PFS" and 95% CI.
- Present a line for each indication (if > 5 patients). Do not display number of patients at risk.




Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

Figure 14.2-1.2

Overall Survival (OS) by Indication (Safety Population)

#### Programming Note:

- Replicate of Figure 14.2-1.1.
- X-axis Label "Overall survival (Months)"
- Y-axix Label "Survival probability (%).
- Present "Median OS" and 95% CI.
- Updated footnote to the following: OS calculated with reference to first dose of Bevacizumab from E-trial.

Figure 14.2-1.3 ation - Exploratory analysis, PFS

Progression Free Survival (PFS) by Indication - Exploratory analysis, PFS with reference to first dose of Bevacizumab from P-trial (Safety Population)

#### Programming Note:

- Replicate of Figure 14.2-1.1.
- Updated footnote to the following: PFS calculated with reference to first dose of Bevacizumab from P-trial.

Figure 14.2-1.4

Overall Survival (OS) by Indication - Exploratory analysis, OS with reference to first dose of Bevacizumab from P-trial (Safety Population)

#### Programming Note:

- Replicate of Figure 14.2-1.1.
- Updated footnote to the following: OS calculated with reference to first dose of Bevacizumab from P-trial.




Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

M025757 -- DELIVERY TYPE -- Table 14.3.1-1.1.1

Page X of Y

# Number (%) of Patients with Adverse Events by Indication, System Organ Class and Preferred Term (Safety Population)

| System Organ Class/<br>Preferred Term | BC<br>(N=X<br>n (% | AND THE RESERVE | nts] | | or PC<br>=XX)<br>(%) [Eve | nts] | CRO<br>(N= | XX) | nts] | RCC<br>(N= | =XX) | nts] | NSC<br>(N= | =XX) | nts] |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Any System Organ Class | XX ( | XXX.X) | [XXX] | XX | (XXX.X) | [XXX] | XX | (XXX.X) | [XXX] | XX | (XXX.X) | [XXX] | XX | (XXX.X) | [XXX] |
| System Organ Class 1 | XX ( | XXX.X) | [XXX] | XX | (XXX.X) | [XXX] | XX | (XXX.X) | [XXX] | XX | (XXX.X) | [XXX] | XX | (XXX.X) | [XXX] |
| Preferred Term 1 | XX ( | XXX.X) | [XXX] | XX | (XXX.X) | [XXX] | XX | (XXX.X) | [XXX] | XX | (XXX.X) | [XXX] | XX | (XXX.X) | [XXX] |
| Preferred Term 2 | XX ( | XXX.X) | [XXX] | XX | (XXX.X) | [XXX] | XX | (XXX.X) | [XXX] | XX | (XXX.X) | [XXX] | XX | (XXX.X) | [XXX] |
| Preferred Term 3 | XX ( | XXX.X) | [XXX] | XX | (XXX.X) | [XXX] | XX | (XXX.X) | [XXX] | XX | (XXX.X) | [XXX] | XX | (XXX.X) | [XXX] |
| (cont.) | XX ( | XXX.X) | [XXX] | XX | (XXX.X) | [XXX] | XX | (XXX.X) | [XXX] | XX | (XXX.X) | [XXX] | XX | (XXX.X) | [XXX] |
| (cont.) | XX ( | XXX.X) | [XXX] | XX | (XXX.X) | [XXX] | XX | (XXX.X) | [XXX] | XX | (XXX.X) | [XXX] | XX | (XXX.X) | [XXX] |

Note: MedDRA version version number>.

A patient with multiple occurrences of an AE is counted only once in each SOC and/or PT.

Source : Listing XXXXXX

<Program Path\Program name.sas> <run on: datetime>

# Programming Note:

- Include all Indications (additional columns), including Total, if possible try to fit all column in 1 page.
- Order the SOC and PT by decreasing frequency.




Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

BMSOP111/F2

Table 14.3.1-1.1.2

Number (%) of Patients with Severe (Grade 3-5) Adverse Events Related to Bevacizumab by Indication,
System Organ Class and Preferred Term
(Safety Population)

# Programming Note:

- Replicate of Table 14.3.1-1.1.1.

Template Author: 
Version 3.0 16AUG2017



Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

M025757 -- DELIVERY TYPE -- Table 14.3.1-1.2.1

Page X of Y

Number (%) of Patients with Adverse Events Related to Bevacizumab by Indication, System Organ Class, Preferred Term and Maximum Severity (Safety Population)

Indication: <indication>

| System Organ Class/<br>Preferred Term | Grade 1<br>(N=XX)<br>n (%) | Grade 2<br>(N=XX)<br>n (%) | Grade 3<br>(N=XX)<br>n (%) | Grade 4<br>(N=XX)<br>n (%) | Grade 5 (N=XX) n (%) | Any Grade<br>(N=XX)<br>n (%) |
|---|---|---|---|---|---|---|
| Any System Organ Class | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| System Organ Class 1 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Preferred Term 1 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Preferred Term 2 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Preferred Term 3 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| System Organ Class 2 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Preferred Term 1 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Preferred Term 2 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| System Organ Class 3 | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |
| Preferred Term 1 (cont.) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) | XX (XXX.X) |

Note: MedDRA version version number>.

A patient with multiple occurrences of an AE is counted only once in each SOC, PT and/or maximum severity.

Source : Listing XXXXXX

<Program Path\Program name.sas> <run on: datetime>

# Programming Note:

- Repeat for each Indication.
- Order the SOC and PT by decreasing frequency.




Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

Table 14.3.1-1.3.1

Number (%) of Patients with Adverse Events Leading to Discontinuation of Bevacizumab by Indication, System Organ Class and Preferred Term
(Safety Population)

# Programming Note:

- Replicate of Table 14.3.1-1.1.1.

Table 14.3.1-1.3.2

Number (%) of Patients with Adverse Events Leading to Discontinuation of Bevacizumab/non-IMP by Indication, System
Organ Class and Preferred Term
(Safety Population)

#### Programming Note:

- Replicate of Table 14.3.1-1.1.1.




Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

Table 14.3.1-1.4.1

Number (%) of Patients with Adverse Events Leading to Discontinuation of Bevacizumab by Indication, System Organ Class, Preferred Term and Maximum Severity (Safety Population)

# Programming Note:

- Replicate of Table 14.3.1-1.2.1.

Table 14.3.1-1.4.2

Number (%) of Patients with Adverse Events Leading to Discontinuation of Bevacizumab/non-IMP by Indication, System Organ Class, Preferred Term and Maximum Severity

(Safety Population)

#### Programming Note:

- Replicate of Table 14.3.1-1.2.1.




Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

M025757 -- DELIVERY TYPE -- Table 14.3.1-1.5.1

Page X of Y

# Number (%) of Patients with Adverse Events of Special Interest (AESI) by Indication, AESI Category and Preferred Term (Safety Population)

| AESI Category/<br>Preferred Term | BC<br>(N=XX)<br>n (%) [Events] | OC or PC<br>(N=XX)<br>n (%) [Events] | CRC<br>(N=XX)<br>n (%) [Events] | RCC (N=XX) n (%) [Events] | NSCLC<br>(N=XX)<br>n (%) [Events] |
|---|---|---|---|---|---|
| Any AESI | xx (xxx.x) [xx | xx (xxx.x) [xx] | xx (xxx.x) [xx] | xx (xxx.x) [xx] | xx (xxx.x) [xx] |
| Hypertension | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] |
| Preferred Term 1 | XX (XXX.X) [XX | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] |
| Preferred Term 2 | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] |
| Preferred Term 3 | XX (XXX.X) [XX | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] |
| (cont.) | XX (XXX.X) [XX | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] |
| (cont.) | XX (XXX.X) [XX | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] | XX (XXX.X) [XX] |

Note: MedDRA version <version number>.

A patient with multiple occurrences of an AE is counted only once in each AESI category and/or PT.

A PT can contribute to more than one AESI category.

Source : Listing XXXXXX

<Program Path\Program name.sas> <run on: datetime>

#### Programming Note:

- Include all Indications (additional columns), including Total, if possible try to fit all column in 1 page.
- List all the AESI categories as presented in the SAP, if there is zero case, please display the AESI with 0 patients.
- AESI category and PT are sorted by decreasing frequency
- SOC will be updated by AESI and PT will be the preferred terms that fall under the AESI category
- A PT can be contributing to more than one AESI category.

 BMSOP111/F2



Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

Table 14.3.1-1.6.1

Number (%) of Patients with Adverse Events of Special Interest (AESI)
by Indication, AESI Category, Preferred Term and
Maximum Severity
(Safety Population)

# Programming Note:

- Replicate of Table 14.3.1-1.2.1.
- Repeat for each Indication and P-trial.
- List all the AESI categories as presented in the SAP, if there is zero case, please display the AESI with 0 patients.
- AESI category and PT are sorted by decreasing frequency
- SOC will be updated by AESI and PT will be the preferred terms that fall under the AESI category
- A PT can be contributing to more than one AESI category.

Table 14.3.1-1.7.1

Number (%) of Patients with Adverse Events Leading to Death by Indication, System Organ Class and Preferred Term (Safety Population)

#### Programming Note:

- Replicate of Table 14.3.1-1.1.1.




Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

Table 14.3.1-1.8.1

Number (%) of Patients with Non-Serious Adverse Events by Indication, System Organ Class and Preferred Term (Incidence ≥ 5% in any Indication)

(Safety Population)

# Programming Note:

- Replicate of Table 14.3.1-1.1.1.




Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

M025757 -- DELIVERY TYPE -- Table 14.3.1-2.1

Page X of Y

Number (%) of Patients with Serious Adverse Events by Indication, System Organ Class and Preferred Term (Safety Population)

Indication: BC

| System Organ Class/<br>Preferred Term | Bevacizumab<br>Total<br>(N=XX) Clopper-Pearson<br>n (%) (95% CI) |
|---|---|
| Any System Organ Class | XX (XXX.X) (XXX.X; XXX.X) |
| System Organ Class 1 | XX (XXX.X) (XXX.X; XXX.X) |
| Preferred Term 1 | XX (XXX.X) (XXX.X; XXX.X) |
| Preferred Term 2 | XX (XXX.X) (XXX.X; XXX.X) |
| Preferred Term 3 | XX (XXX.X) (XXX.X; XXX.X) |
| (cont.) | XX (XXX.X) (XXX.X; XXX.X) |
| (cont.) | XX (XXX.X) (XXX.X; XXX.X) |

Note: MedDRA version version number>.

A patient with multiple occurrences of an AE is counted only once in each SOC and/or PT.

Source : Listing XXXXXX

<Program Path\Program name.sas> <run on: datetime>

# Programming Note:

- Repeat for each Indication including Total.
- SOC category and PT are sorted by decreasing frequency




Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

Table 14.3.1-2.2

Number (%) of Patients with Severe (Grade 3-5) Adverse Events Related to Bevacizumab by Indication,
System Organ Class and Preferred Term
(Safety Population)

# Programming Note:

- Replicate of Table 14.3.1-2.1.




Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

M025757 -- DELIVERY TYPE --

Page X of Y

# Table 14.3.1-4.1

Cause of Death and Relationship of Death to Study Treatment by Indication (Safety Population)

P-trial: Overall

| | BC<br>(N=XX)<br>n (%) | (N | or PC<br>=XX)<br>(%) | CRC<br>(N=XX)<br>n (%) | RCC<br>(N=XX)<br>n (%) | NSCLC<br>(N=XX)<br>n (%) | GBM<br>(N=XX)<br>n (%) |
|---|---|---|---|---|---|---|---|
| No of patients who died | XXX (X | XX.X) XX | x (xxx.x) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) |
| Cause of death* | | | | | | | |
| Progressive disease | XXX (X | XX.X) XX | X (XXX.X) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) |
| Adverse event | XXX (X | XX.X) XX | X (XXX.X) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) |
| Other | XXX (X | XX.X) XX | X (XXX.X) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) |
| Relationship of death to Be | vacizumab* | | | | | | |
| Related | XXX (X | XX.X) XX | X (XXX.X) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) |
| Unrelated | XXX (X | XX.X) XX | X (XXX.X) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) |
| Relationship of death to Ot | her Non-IM | P* | | | | | |
| Related | XXX (X | XX.X) XX | X (XXX.X) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) |
| Unrelated | XXX (X | XX.X) XX | X (XXX.X) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) | XXX (XXX.X) |

Note: \* Percentages are calculated from the number of patients who died within the indication considered.

Source : Listing XXXXXX

<Program Path\Program name.sas> <run on: datetime>

# Programming Note:

- Include all Indications (additional columns), including Total, if possible, fit all column in the same page.

Template Author:  BMSOP111/F2

Version 3.0 16AUG2017



**Statistical Analysis Plan:** Final version 3.0 / 18-FEB-2019

Page X of Y

M025757 -- DELIVERY TYPE -- Listing 16.2.1-1

End of Treatment/Study
(All Patients Population)

Indication: XXXX P-trial: XXXXX

Non-IMP: XXXXXXX

| Country/<br>Center/<br>Patient | Age/ Safety<br>Sex Pop.? | First dose date/<br>Last dose date<br>(day) [a] | Visit | Days since initial treat. in P-trial [c] | | Reason for discontinuation, specify | Date consent withdrawn | Observation time (months)[b] |
|---|---|---|---|---|---|---|---|---|
| XXXX/XXXX/XXXX | XX/X Yes | DDMMMYYYY/ | ЕоТ | X | | Adverse Event | | |
| | | DDMMMMYYYY (XXX) | EoS | XX | No | Other, XXXXX | | XX.X* |
| XXXX/XXXX/XXXX | XX/X Yes | DDMMMYYYY/<br>DDMMMMYYYY (XXX) | EoT | XX | | Withdrawal of consent | DDMMMYYYY | |
| | | DDIMENTITI (IIIII) | EoS | XX | Yes | | | XX.X |
| XXXX/XXXX/XXXX | XX/X No | | EoS | | No | XXXXX | DDMMMYYYY | |

<sup>[</sup>a] First and last dose date of Bevacizumab treatment. Day is relative to the first dose date of treatment in the E-trial.

<sup>[</sup>b] Observation time is calculated as the time to safety follow-up visit from first bev. admin in E-trial.

<sup>[</sup>c] Days since initial treatment in P-trial is relative to the first dose date of treatment (Bevacizumab) in the P-trial. \* censored.

<sup>&</sup>lt;Program Path\Program name.sas> <run on: datetime>



**Statistical Analysis Plan:** Final version 3.0 / 18-FEB-2019

Page X of Y

M025757 -- DELIVERY TYPE --

Listing 16.2.2-1 Protocol Deviations (All Patients Population)

Indication: XXXX; P-trial: XXXXX

Non-IMP: XXXXXXX

| Country/<br>Center/<br>Patient | Age/<br>Sex | Date of Protocol<br>Deviation (day) [a] | Protocol Deviation<br>Category | n<br>Protocol Deviation Description | Included in summary? [b] |
|---|---|---|---|---|---|
| XXXX/XXXX/XXXX | XX/X | DDMMMMYYYY (XXX)<br>DDMMMMYYYY (XXX) | XXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXX<br>XXXXXXX |
| XXXX/XXXX/XXXX | XX/X | DDMMMMYYYY (XXX) | XXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |

<sup>[</sup>a] Day is relative to the first dose date of treatment in the E-trial.

<Program Path\Program name.sas> <run on: datetime>

 BMSOP111/F2

<sup>[</sup>b] Major protocol deviations from inclusion criteria 2 and 3, exclusion criteria 8 and 10 or anything else that is a major protocol deviation potentially impacting the primary endpoint (AE grade >=3 rates) or put patient at risk.



**Statistical Analysis Plan:** Final version 3.0 / 18-FEB-2019

M025757 -- DELIVERY TYPE -- Listing 16.2.4-1.1

Page X of Y

# Demographics and Baseline Characteristics (All Patients Population)

Indication: XXXX P-trial: XXXXX

Non-IMP: XXXXXXX

| Country/<br>Center/<br>Patient | Age/<br>Sex | Date of<br>birth | Tumour Type | Indication | | Baseline<br>Weight (kg) |
|---|---|---|---|---|---|---|
| XXXX/XXXX/XXXX<br>XXXX/XXXX/XXXX | XX/X<br>XX/X | DDMMMYYYY | XXXXX | xxxxxxx | : | XX.X |

Note: Baseline is defined as the Cycle for which the first dose of Bevacizumab was administered.

<Program Path\Program name.sas> <run on: datetime>

 BMSOP111/F2



Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

Page X of Y

M025757

-- DELIVERY TYPE --Listing 16.2.4-1.2 P-trial Information (All Patients Population)

Indication: XXXXX P-trial: XXXXX

| | | Ве | evacizumab | | | |
|---|---|---|---|---|---|---|
| Country/<br>Center/<br>Patient | Age/Site<br>Sex Nb. | | Date of last<br>dose (day) [a] | Dose Regimen on<br>P-trial | Continued with other Ptrial IMP? | O-<br>Other IMPs from P-trial |
| XXXX/XXXX/XXXX | XX/X XXXX | DDMMMYYYY | DDMMMYYYY<br>(XXX) | 7.5 mg/kg IV<br>every 21 days | Yes | Interferon alpha-2a |
| XXXX/XXXX/XXXX | XX/X XXXX | | , | 1 1 | | |

 BMSOP111/F2

<sup>[</sup>a] Day is relative to the first dose date of Bevacizumab in the P-trial.

<sup>&</sup>lt;Program Path\Program name.sas> <run on: datetime>



**Statistical Analysis Plan:** Final version 3.0 / 18-FEB-2019

Page X of Y

M025757

-- DELIVERY TYPE --Listing 16.2.4-2 Pregnancy Test (All Patients Population)

Indication: XXXX; P-trial: XXXXX

Non-IMP: XXXXXXX

| Country/<br>Center/ | Age/ | | Pregnancy test | | | Date (day) | of | |
|---|---|---|---|---|---|---|---|---|
| Patient | Sex | Visit | done? | Reasor | n not done | sample | | Result |
| XXXX/XXXX/XXXX | XX/X | Screening | Yes | | | DDMMMYYYY | (-XX) | Negative |
| XXXX/XXXX/XXXX | XX/X | Screening | No | Other, | XXXXXX | | | |

Note: Day is relative to the first dose of treatment in the E-trial.

<Program Path\Program name.sas> <run on: datetime>

 BMSOP111/F2



Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

Page X of Y

M025757 -- DELIVERY TYPE -- Listing 16.2.5-1.1

Administration of Bevacizumab (Safety Population)

Indication: XXXX P-trial: XXXXX

Non-IMP: XXXXXXX

| Country/<br>Center/<br>Patient | Age/<br>Sex | Baseline<br>weight<br>(kg) | Cycle | Date (day)<br>dose<br>administere | ed | Dose (mg) administered | Weight<br>(kg) | Dose<br>(mg/kg) | Compliance (%) | Reason dose not given, specify | Flag* |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXX/XXXX/XXXX | XX/X | XX.X<br>XX.X | Cycle 1<br>Cycle 2<br>Cycle 3<br>Overall | DDMMMYYYY | . , | XXX.X<br>XXX.X | XX.X<br>XX.X | XX.X<br>XX.X<br>XX.X<br>XX.X | XX.X<br>XX.X<br>XX.X | Other, XXXXX | * |
| XXXX/XXXX/XXXX | XX/X | | Cycle 1 | | | | | | | | |

Note: Day is relative to the first dose of treatment in the E-trial.

<Program Path\Program name.sas> <run on: datetime>

 BMSOP111/F2

<sup>\*</sup> Dose is reduced for reasons other than a >10% change (loss or gain) in weight from baseline.



Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

Page X of Y

M025757 -- DELIVERY TYPE -Listing 16.2.5-1.2
Administration of non-IMP Treatment

Administration of non-IMP Treatment (Safety Population)

Indication: XXXX P-trial: XXXXX

XXXX/XXXX/XXXX XX/X Cycle 1

Non-IMP: XXXXXXX

| Country/<br>Center/<br>Patient | Age/<br>Sex | Cycle | Drug name | Date (day) dose<br>administered/ Last<br>dose date (day) in<br>cycle [a] | , , | fadmin.as | s Percentage | Reason dose modified/<br>not given, specify<br>[b] |
|---|---|---|---|---|---|---|---|---|
| XXXX/XXXX/XXXX | XX/X | Cycle 1 | xxxxxxxxx | DDMMMYYYY (1)/ DDMMMYYYY (XX) DDMMMYYYY (1)/ DDMMMYYYY (XX) | XXX.X (XX)/<br>2 dose<br>XXX.X (XX)/<br>1 dose | No<br>Yes | 85% | XXXXXXXX |
| | | Cycle 2 | | DDMMMYYYY (XX) /<br>DDMMMYYYY (XX) | XXX.X (XX)/<br>2 dose | XXX | | |
| | | Cycle 3 | | DDMMMYYYY (XX) /<br>DDMMMYYYY (XX) | | No | 0% | Other, XXXXX |
| | | Cycle 4 | XXXXXXXX | DDMMMYYYY (XX) | | | | Adverse Event |

Note: Day is relative to the first dose of treatment in the E-trial.

<Program Path\Program name.sas> <run on: datetime>


 BMSOP111/F2

<sup>[</sup>a] If the non-IMP administration was discontinued, the date (day) of last dose is presented

<sup>[</sup>b] If the non-IMP administration was discontinued, the reason the non-IMP were discontinued is displayed.



Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

Page X of Y

M025757 -- DELIVERY TYPE -Listing 16.2.5-2
Duration of exposure to Bevacizumab

(Safety Population)

Indication: XXXX P-trial: XXXXX

Non-IMP: XXXXXXX

| Country/<br>Center/<br>Patient | Age/<br>Sex | Treatment duration of Bev.(E-trial) (months) [a] | Treatment duration of Bev. (overall) (months) [b] | Approximate number of cycles (overall) [c] |
|---|---|---|---|---|
| XXXX/XXXX/XXXX | XX/X | XX.X | XX.X | XX.X |
| XXXX/XXXX/XXXX | XX/X | XX.X | XX.X | XX.X |
| XXXX/XXXX/XXXX | XX/X | XX.X | XX.X | xx.x |

Note: Day is relative to the first dose of treatment in the E-trial.

[a] Treatment Duration of Bev. (E-trial) = [(Date of last dose of Bev. in E-trial - Date of first dose of Bev. in E-trial) + 1]/ 30.4375.

[b] Treatment Duration of Bev. (overall) = [(Date of last dose of Bev. in E-trial - Date of first dose of Bev. in P-trial) + 1]/30.4375.

[c] Approximate number of Cycles (overall) = [(Date of last dose of Bev. in E-trial - Date of first dose of Bev. in P-trial) + 1] / (number of days in a cycle).

<Program Path\Program name.sas> <run on: datetime>

M025757 -- DELIVERY TYPE -- Page X of Y

Listing 16.2.6-1.1 Time to Event (Safety Population)

Indication: XXXX; P-trial: XXXXX

Non-IMP: XXXXXXX

Template Author:  BMSOP111/F2

Version 3.0 16AUG2017



**Statistical Analysis Plan:** Final version 3.0 / 18-FEB-2019

| Country/<br>Center/<br>Patient | Age/<br>Sex | Progression Free<br>Survival (mths.)<br>[1] | Overall Survival (mths.) [1] | Progression Free<br>Survival (mths.) -<br>Exploratory analysis<br>[2] | Overall Survival (mths.) - Exploratory analysis [2] |
|---|---|---|---|---|---|
| XXXX/XXXX/XXXX | XX/X | XXX | XXX | XXX | XXX |
| XXXX/XXXX/XXXX | XX/X | XXX | XXX* | XXX | XXX* |
| XXXX/XXXX/XXXX | XX/X | XXX | XXX | XXX | XXX |
| XXXX/XXXX/XXXX | XX/X | XXX | XXX | XXX | XXX |
| XXXX/XXXX/XXXX | XX/X | XXX* | XXX | XXX* | XXX |
| XXXX/XXXX/XXXX | XX/X | XXX | XXX* | XXX | XXX |
| (cont.) | | | | | |

Note: Time to event is relative to the first dose of treatment in the E-trial (or in the P-trial for the exploratory analysis).


 BMSOP111/F2

<sup>[1]</sup> Progression Free Survival/Overall Survival calculated with reference to first dose of Bevacizumab from E-trial.

<sup>[2]</sup> Progression Free Survival/Overall Survival calculated with reference to first dose of Bevacizumab from P-trial. 1 month=30.4375 days.

<sup>\*</sup> censored.

<sup>&</sup>lt;Program Path\Program name.sas> <run on: datetime>



Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

Page X of Y

M025757 -- DELIVERY TYPE --

Listing 16.2.6-1.2
Progression Assessment
(Safety Population)

Indication: XXXX; P-trial: XXXXX

Non-IMP: XXXXXXX

| Country/<br>Center/<br>Patient | Age/<br>Sex | Cycle | Date (day) of assessment | Disease<br>progression? | Date (day) of progression | How progression was assessed? | RECIST<br>version |
|---|---|---|---|---|---|---|---|
| XXXX/XXXX/XXXX | XX/X | Cvcle 1 | DDMMMYYYY (XXX) | No | | Clinical Assessment | |
| | ΛΛ/ Λ | Cycle 1 | DDMMMYYYY (XXX) | No | | Clinical Assessment | |
| | | Cycle 3 | DDMMMYYYY (XXX) | ND | | CIIIIICAI ASSESSMENC | |
| | | 4 | , , | | | Dadialanias Assassmen | - 171 0 |
| | | Cycle 4 | DDMMMYYYY (XXX) | Yes | DDMMMYYYY (XXX) | Radiological Assessmen | VI.U |
| XXXX/XXXX/XXXX | XX/X | | | | | | |

Note: Day is relative to the first dose of treatment in the E-trial.

RECIST=Response Evaluation Criteria in Solid Tumours; ND=Not Done; NE=Assessment not scheduled at this visit. Assessments for progression disease done as per the local standard, although it is recommended to continue using the same methods as in the P-trial.

<Program Path\Program name.sas> <run on: datetime>

 BMSOP111/F2



Statistical Analysis Plan: Final version 3.0 / 18-FEB-2019

M025757 -- DELIVERY TYPE -- Listing 16.2.7-1

Adverse Events (Safety Population)

Indication: XXXX P-trial: XXXXX

Non-IMP: XXXXXXX

| Country/<br>Center/<br>Patient | Age/<br>Sex | Adverse Event (REPORTED)/<br>Preferred Term/<br>System Organ Class | Start date | _ | Days since last treat. in E-trial [a] | Duration<br>(days)/<br>Severity*/<br>SAE?/AESI? | Related to<br>Bevacizumab/<br>Non-IMP | Action Taken<br>Concomitant<br>med non<br>drug?/<br>Outcome | Action<br>Taken with<br>Bevacizumab<br>/Non-IMP |
|---|---|---|---|---|---|---|---|---|---|
| XXXX/XXXX/XXXX | XX/X | XXXXXXXX/<br>XXXXXXXXX<br>XXXXXXXXX/<br>XXXXXXXX | | (XXX) | -XXX | XXX/ Grade 1 (4.0)/ No/No XXX/ Grade 5 (4.1)/ | Not Rel./ | Yes/<br>No/<br>Resolved<br>None/<br>Yes/ | Inter./ Disc. None/ Adjusted |
| xxxx/xxxx/xxxx | XX/X | ************************************** | DDMMMYYYY<br>DDMMMYYYY | | -xx | Yes/Yes XXX/ Grade 1 (4.0)/ No/Yes | Rel./<br>Not Rel. | Yes/<br>No/<br>Unres. | Disc./<br>Non |

Note: Day is relative to the first dose of treatment in the E-trial. Study day will be derived based on imputed dates.

\* version of the NCI-CTCAE used is displayed in parenthesis. \$ Ongoing from P-trial.

MedDRA version <x.x>.

[a] Days since last treatment in E-trial is relative to the last dose date of treatment (Bevacizumab) in the E-trial. Abbreviations: Disc=Discontinued; Inter=Interrupted; Rel=Related; Unres=Unresolved/Ongoing (at Safety Follow Up).

<Program Path\Program name.sas> <run on: datetime>

Page X of Y



**Statistical Analysis Plan:** Final version 3.0 / 18-FEB-2019

Page X of Y

M025757 -- DELIVERY TYPE --

Listing 16.2.7-2
All Deaths
(Safety Population)

Indication: XXXX P-trial: XXXXX

Non-IMP: XXXXXXX

| Country/<br>Center/<br>Patient | Age/<br>Sex | Cause of death | Adverse<br>event or<br>prefered<br>term (if<br>other) | Date (day)<br>death | of | Days since<br>last treat.<br>E-trial [a] | in Related to<br>Bevacizumab | | AE/SAE reported? |
|---|---|---|---|---|---|---|---|---|---|
| XXXX/XXXX/XXXX | XX/X | Adverse Event | XXXXXXXXXX | DDMMMYYYY | (XXX) | -XXX | Related | Not related | Yes |
| XXXX/XXXX/XXXX | XX/X | Other | XXXXXXXXXX | DDMMMYYYY | (XXX) | -XXXX | Not related | Not related | No |
| XXXX/XXXX/XXXX | XX/X | Progressive disease | | DDMMMYYYY | (XXX) | -xxx | Not related | Not related | No |

Note: Day is relative to the first dose of treatment in the E-trial.

 BMSOP111/F2

<sup>[</sup>a] Days since last treatment in E-trial is relative to the last dose date of treatment (Bevacizumab) in the E-trial.

<sup>&</sup>lt;Program Path\Program name.sas> <run on: datetime>



Sponsor: ROCHE
Protocol: MO25757
Statistical Analysis Plan:

Final version 3.0 / 18-FEB-2019

# 12.2 Imputation of partial dates

With regards to missing start and stop date for AEs the following imputation rules will be followed.

# Stop dates:

- o If the AE is not ongoing and the stop date is partial (day or day/month missing), the stop date will be imputed by the last day of the month if the day is missing, the 31<sup>st</sup> of December if the day and month is missing or the date of death (if occurred on the same year or same month and year as the stop date), whichever date occurred first.
- If the AE is not ongoing and the stop date is missing, the stop date will be imputed by the start date (if complete), by the last day of the month the AE started (if only day is missing), by the 31<sup>st</sup> of December of the year the AE started (if the day and month are missing) and by the first dose of treatment (if the start date is missing)
- Start dates: once the stop dates have been imputed as above the following rules will be used:
  - If the start date is missing it will be imputed by the date of the first dose of treatment
  - o If the day is missing it will be imputed by the last day of the month
  - If the day and month are missing they will be imputed by the 31<sup>st</sup> of December
  - o If the start date once imputed is after the stop date, the start date will be imputed with the stop date.
  - If the start date once imputed is after the date of death, the start date will be imputed with date of death.